CLINICAL TRIAL: NCT07213050
Title: Percutaneous Thermal Ablation (Radiofrequency and Microwave) in the Treatment of Anterior Abdominal Wall Masses: An Evaluation of Efficacy and Safety.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MOHAMED ALI IBRAHIM ABOLOYOUN SAYED, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Percutaneous Thermal Ablation
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Anterior Abdominal Wall Masses
MeSH Terms: interventions — Microwaves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Active Comparator): Patients with biopsy-proven metastases to the anterior abdominal wall (e.g.,from colorectal, breast, ovarian cancer)
  Interventions: Procedure: Radiofrequency; Procedure: Microwave

INTERVENTIONS:
Procedure: Radiofrequency — achieve a target temperature of 90-110°C for 4-12 minutes, ensuring an ablative margin of at least 0.5-1.0 cm around the tumor.
Procedure: Microwave — Antennas will be placed under imaging guidance, and ablation will be performed for 5-10 minutes per antenna activation to achieve the desired margin.

SUMMARY:
The anterior abdominal wall is a common site for metastatic deposits (e.g., from colorectal, ovarian, or hepatocellular carcinoma), desmoid tumors (aggressive fibromatosis), and endometriomas. Surgical resection has been the traditional standard of care. However, surgery in this region can be complex due to the proximity of vital structures, the need for large tissue resection, and high recurrence rates. Furthermore, patients often present with significant comorbidities or have recurrent disease after previous surgeries, making them poor surgical candidates While established in organs like the liver and lungs, their application specifically for abdominal wall lesions is a growing and evidence-supported field that warrants further systematic study to standardize protocols and confirm long-term outcomes.

Percutaneous thermal ablation, including microwave ablation (MWA) and radiofrequency ablation (RFA), is an increasingly used minimally invasive treatment for anterior abdominal wall lesions such as metastatic tumors and benign lesions like abdominal wall endometriosis. These techniques deliver thermal energy through percutaneous probes to induce coagulative necrosis, offering an effective alternative to surgery with lower morbidity and shorter recovery times.

RFA uses high-frequency electrical currents to generate heat and ablate tumors. It is well established for treating abdominal wall recurrences, particularly from colorectal cancer, with effective local control and symptom relief.

Ultrasound-guided MWA has demonstrated excellent safety and efficacy for abdominal wall lesions. Studies report significant lesion volume reduction, pain relief, and low complication rates in patients with abdominal wall endometriosis and metastases. The ability to visualize the ablation zone in real-time with ultrasound enhances precision and protects adjacent structures.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with biopsy-proven metastases to the anterior abdominal wall (e.g., from colorectal, breast, ovarian cancer). 2. Patients with biopsy-proven desmoid tumors (aggressive fibromatosis). 3. Patients with symptomatic abdominal wall endometriomas. 4. Lesion size ≤ 5 cm in greatest diameter. 5. Patients deemed unfit for surgery due to comorbidities, or who refuse surgical intervention. 6. Platelet count > 50,000/µL and INR < 1.5.

Exclusion Criteria:

* 1. Uncorrectable coagulopathy. 2. Lesion size > 5 cm. 3. Unlimited diffuse peritoneal carcinomatosis. 4. Skin or bowel wall involvement with no safe percutaneous pathway for ablation (as determined on pre-procedural CT) 5. Life expectancy < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success | baseline
  complete coverage of the target lesion by the ablation zone with an adequate margin on the immediate post-procedure CT scan